CLINICAL TRIAL: NCT02267564
Title: Medial Patellofemoral Ligament (MPFL) Reconstruction With or Without Tibial Tubercle Transfer for Recurrent Patellar Instability
Brief Title: MPFL Reconstruction With or Without Tibial Tubercle Transfer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yu Jiakuo (Other)
Responsible Party: Sponsor-Investigator, Yu Jiakuo, Professor, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014099
Record Dates: First submitted 2014-09-28; First posted 2014-10-17 (Estimated); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Patellar Dislocation
Keywords: patellar dislocation; medial patellofemoral ligament; tibial tubercle transfer
MeSH Terms: conditions — Patellar Dislocation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MPFLR without tibial tubercle transfer (Experimental): Patients with patellar instability undergo MPFL reconstruction without tibial tubercle transfer.
  Interventions: Procedure: MPFL reconstruction; Procedure: tibial tubercle transfer
- MPFLR with tibial tubercle transfer (Active Comparator): Patients with patellar instability undergo MPFL reconstruction with tibial tubercle transfer.
  Interventions: Procedure: MPFL reconstruction; Procedure: tibial tubercle transfer

INTERVENTIONS:
Procedure: MPFL reconstruction — to correct patellar dislocation with medial patellofemoral ligament reconstruction
Procedure: tibial tubercle transfer — to correct patellar dislocation with tibial tubercle medial transfer

SUMMARY:
This study aims to compare the clinical outcome of Medial PatelloFemoral Ligament (MPFL) reconstruction with and without tibial tubercle transfer for recurrent patellar dislocation.

DETAILED DESCRIPTION:
70 patients with recurrent patellar instability were randomly assigned to undergo MPFL reconstruction with or without tibial tubercle transfer. Follow-ups were performed at 12 and 24 months postoperatively, and computed tomography (CT) was performed immediately after the operation and at follow-up. The knee function was evaluated preoperatively and at 2 years postoperatively using Lysholm,Tegner and Kujala scales. Redislocation or multiple episodes of patellar instability were considered failures.

ELIGIBILITY:
Inclusion Criteria:

* recurrent patellar dislocation or instability,patients with TT-TG value equal to or greater than 20 mm,patients with closed epiphyseal plate

TT-TG：Two lines drawn perpendicular to posterior bicondylar line, one line through middle of the trochlear groove(TG) and the second through tibial tuberosity (TT). Distance between the lines is measured.

Exclusion Criteria:

* bilateral patellar dislocation, a previous surgery in the involved leg,patients with open epiphyseal plate,patients with severe trochlear dysplasia

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Lysholm score of the knee | two years
  Lysholm score of the knee was evaluated preoperatively and at 2 years post operation .
  Scale name:score
Tegner score of the knee | two years
  Tegner score of the knee was evaluated preoperatively and at 2 years post operation .
  Scale name:score
Kujala score of the knee | two years
  Kujala score of the knee was evaluated preoperatively and at 2 years post operation .

SECONDARY OUTCOMES:
CT images of the knee | two years
  CT was performed immediately after the operation and at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Kuo Yu, Doctor, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China